CLINICAL TRIAL: NCT06726993
Title: Comparison of Restricted Kinematic Alignment Versus Unrestricted Kinematic Alignment in Primary Total Knee Arthroplasty:- Randomized Controlled Trial
Brief Title: Comparison of Restricted Versus Unrestricted Kinematic Alignment in 1ry TKA
Acronym: rKA-KA-TKA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sohibe Abdulazeem Ghietah Hussein, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2024-100320
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis (OA) of the Knee; Total Knee Anthroplasty
Keywords: Total knee arthroplasty; TKA; Total knee replacement; TKR; Restricted kinematic alignment; rKA; Kinematic alignment; KA; Unrestricted kinematic alignment
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unrestricted kinematic alignment (Experimental): reproducing the constitutional tibiofemoral tridimensional alignment and knee laxity. It is almost a pure bone procedure with only exceptional collateral ligament release, which has been shown to reliably position knee components.
  Interventions: Procedure: Total knee arthroplasty
- Restricted kinematic alignment (Experimental): reproducing patient's constitutional knee anatomy within a safe range while avoiding extreme or pathological anatomies that have been demonstrated to exist.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Total knee arthroplasty (TKA) is a common orthopaedic surgery that involves replacing the articular surfaces (femoral condyles and tibial plateau) of the knee joint with smooth metal and highly cross-linked polyethylene plastic
  Other Names: Total knee replacement

SUMMARY:
Knee osteoarthritis is a growing socioeconomic burden because of the ageing and obesity. By 2030, the majority of individuals undergoing knee arthroplasty in USA will be those younger than 65 years, with up to 1 million achieved annually.

The definitive treatment for knee joint degeneration is total knee arthroplasty.

DETAILED DESCRIPTION:
Furthermore, the commonest technique is neutral mechanical alignment total knee arthroplasty. Latest studies have revealed that the mechanical alignment technique repeatedly causing substantial anatomical alterations with a widespread of complex collateral ligament imbalances, which are not repairable by collateral ligament release. Consequently, the total knee arthroplasty individuals walk with an abnormal gait, and they do not experience a normal knee joint. This may be one of the causes that up to 20% of total knee arthroplasty individuals are disappointed, and over 50% may have remaining symptoms.

Consequently, the conventional mechanical alignment technique has been recently challenged by a new alternative technique, namely unrestricted kinematic alignment proposed by Howell, as a possible solution to the high dissatisfaction following total knee arthroplasty, aiming at reproducing the constitutional tibiofemoral tridimensional alignment and knee laxity. It is almost a pure bone procedure with only exceptional collateral ligament release, which has been shown to reliably position knee components.

The restricted kinematic alignment protocol suggested by Vendittoli has been developed as an alternative to the unrestricted kinematic alignment for patients with an outlier or atypical knee anatomy. The restricted kinematic alignment is founded on five principles: hip-knee-ankle angle should be maintained within ± 3° postoperatively; a limitation to a maximum of 5° for lateral distal femoral angle and medial proximal tibial angle may be considered; restoration of collateral ligament balance should be achieved without the gap balancing technique; native femoral anatomy preservation is suggested over tibial one to maintain knee biomechanics; resurface resection must be accomplished on the unworn side with a thickness equivalent to the width of the implant;cut fine-tuning may be sought at the worn side.

ELIGIBILITY:
Inclusion Criteria:

-Patients suffered from end stage knee osteoarthritis of grade four according to Kellgren-Lawrence classification in at least one of the three knee compartments, who have an osteoarthritic knees of varus Coronal Plane Alignment of the Knee classification

Exclusion Criteria:

1. Any valgus malalignment of the knee joint.
2. Malalignment more than 10° or less than 3° varus of knee joint.
3. Ligamentous laxity of the affected knee (medial or lateral collateral ligaments)
4. any tumors or secondary neoplasia diseases
5. Knee joint infection
6. severe cardiopulmonary dysfunction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Oxoford knee score | 12 months
  The Oxford Knee Score is a 12-item patient-reported outcomes specifically designed and developed to assess function and pain after total knee replacement arthroplasty. It is short, reproducible, valid and sensitive to clinically important changes.
  Score each question from 0 to 4 with 4 being the best outcome. This method, when summed, produces overall scores running from 0 to 48 with 48 being the best outcome

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 24 months
  The Knee Injury and Osteoarthritis Outcome Score is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury. The questionnaire is self-administered and assesses five outcomes: pain(9 items), symptoms(7 items), activities of daily living(17 items), sport and recreation function(5 items), and knee-related quality of life (4 items). The questionnaire meets basic criteria of outcome measures and can be used to evaluate the course of knee injury and treatment outcome.
  A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included.
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Forgotten Joint Score | 24 months
  The Forgotten Joint Score was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. This questionnaire shows its strengths in patients with a good level of knee function and a low pain level. It has been designed specifically to reduce ceiling effects commonly associated with many patients reported outcome measures in this patient group, e.g. when assessing short- to mid-term results in total knee arthroplasty patients.
  Every question is scored 1 (never) to 5 (mostly) according to the selected response categories. Thus, the raw score ranges from 12 to 60. The raw score is linearly transformed to a 0-100 scale and then reversed to obtain the final score.
  Final score = 100 - ((sum(item01 to item12) - 12)/48*100) For the final 'Forgotten Joint Score -12' a high score indicates good outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sohibe A Ghietah, Specialist, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Howell SM HM. Kinematic alignment in TKA: definition, surgical technique, and challenging cases.. Orthopedic Knowledge Online. 2012; 10(7).
- [Background] Risitano S, Cacciola G, Sabatini L, Capella M, Bosco F, Giustra F, Masse A, Vaishya R. Restricted kinematic alignment in primary total knee arthroplasty: A systematic review of radiographic and clinical data. J Orthop. 2022 Jul 2;33:37-43. doi: 10.1016/j.jor.2022.06.014. eCollection 2022 Sep-Oct. PMID 35812351
- [Background] Albishi W, AbuDujain NM, Arafah O, Alshaygy IS, Aldosari ZA, Alhuqbani MN, Alangari SM. Cross-cultural adaptation, validity and reliability of the Arabic version of the Forgotten Joint Score for knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2023 Oct;31(10):4312-4318. doi: 10.1007/s00167-023-07484-y. Epub 2023 Jun 17. PMID 37329371
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Almangoush A, Herrington L, Attia I, Jones R, Aldawoudy A, Abdul Aziz A, Waley A. Cross-cultural adaptation, reliability, internal consistency and validation of the Arabic version of the knee injury and osteoarthritis outcome score (KOOS) for Egyptian people with knee injuries. Osteoarthritis Cartilage. 2013 Dec;21(12):1855-64. doi: 10.1016/j.joca.2013.09.010. Epub 2013 Oct 2. PMID 24095836
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Ahmed KM, Said HG, Ramadan EKA, Abd El-Radi M, El-Assal MA. Arabic translation and validation of three knee scores, Lysholm Knee Score (LKS), Oxford Knee Score (OKS), and International Knee Documentation Committee Subjective Knee Form (IKDC). SICOT J. 2019;5:6. doi: 10.1051/sicotj/2018054. Epub 2019 Mar 8. PMID 30848244
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955
- [Background] MacDessi SJ, Griffiths-Jones W, Harris IA, Bellemans J, Chen DB. Coronal Plane Alignment of the Knee (CPAK) classification. Bone Joint J. 2021 Feb;103-B(2):329-337. doi: 10.1302/0301-620X.103B2.BJJ-2020-1050.R1. PMID 33517740
- [Background] Vendittoli PA, Martinov S, Blakeney WG. Restricted Kinematic Alignment, the Fundamentals, and Clinical Applications. Front Surg. 2021 Jul 20;8:697020. doi: 10.3389/fsurg.2021.697020. eCollection 2021. PMID 34355018
- [Background] Hutt JR, LeBlanc MA, Masse V, Lavigne M, Vendittoli PA. Kinematic TKA using navigation: Surgical technique and initial results. Orthop Traumatol Surg Res. 2016 Feb;102(1):99-104. doi: 10.1016/j.otsr.2015.11.010. Epub 2016 Jan 6. PMID 26776100
- [Background] Ranawat AS, Ranawat CS, Elkus M, Rasquinha VJ, Rossi R, Babhulkar S. Total knee arthroplasty for severe valgus deformity. J Bone Joint Surg Am. 2005 Sep;87 Suppl 1(Pt 2):271-84. doi: 10.2106/JBJS.E.00308. PMID 16140800
- [Background] Howell SM, Howell SJ, Hull ML. Assessment of the radii of the medial and lateral femoral condyles in varus and valgus knees with osteoarthritis. J Bone Joint Surg Am. 2010 Jan;92(1):98-104. doi: 10.2106/JBJS.H.01566. PMID 20048101
- [Background] Bellemans J, Colyn W, Vandenneucker H, Victor J. The Chitranjan Ranawat award: is neutral mechanical alignment normal for all patients? The concept of constitutional varus. Clin Orthop Relat Res. 2012 Jan;470(1):45-53. doi: 10.1007/s11999-011-1936-5. PMID 21656315
- [Background] Nam D, Nunley RM, Barrack RL. Patient dissatisfaction following total knee replacement: a growing concern? Bone Joint J. 2014 Nov;96-B(11 Supple A):96-100. doi: 10.1302/0301-620X.96B11.34152. PMID 25381418
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Collins M, Lavigne M, Girard J, Vendittoli PA. Joint perception after hip or knee replacement surgery. Orthop Traumatol Surg Res. 2012 May;98(3):275-80. doi: 10.1016/j.otsr.2011.08.021. Epub 2012 Mar 28. PMID 22459101
- [Background] Blakeney W, Clement J, Desmeules F, Hagemeister N, Riviere C, Vendittoli PA. Kinematic alignment in total knee arthroplasty better reproduces normal gait than mechanical alignment. Knee Surg Sports Traumatol Arthrosc. 2019 May;27(5):1410-1417. doi: 10.1007/s00167-018-5174-1. Epub 2018 Oct 1. PMID 30276435
- [Background] Almaawi AM, Hutt JRB, Masse V, Lavigne M, Vendittoli PA. The Impact of Mechanical and Restricted Kinematic Alignment on Knee Anatomy in Total Knee Arthroplasty. J Arthroplasty. 2017 Jul;32(7):2133-2140. doi: 10.1016/j.arth.2017.02.028. Epub 2017 Feb 20. PMID 28302462
- [Background] Cherian JJ, Kapadia BH, Banerjee S, Jauregui JJ, Issa K, Mont MA. Mechanical, Anatomical, and Kinematic Axis in TKA: Concepts and Practical Applications. Curr Rev Musculoskelet Med. 2014 Jun;7(2):89-95. doi: 10.1007/s12178-014-9218-y. PMID 24671469
- [Background] Riviere C, Iranpour F, Harris S, Auvinet E, Aframian A, Chabrand P, Cobb J. The kinematic alignment technique for TKA reliably aligns the femoral component with the cylindrical axis. Orthop Traumatol Surg Res. 2017 Nov;103(7):1069-1073. doi: 10.1016/j.otsr.2017.06.016. Epub 2017 Sep 1. PMID 28870873